CLINICAL TRIAL: NCT04098029
Title: The Protocol of Estimation of the Safety and Efficiency of the Method of Transfusion of UCB Hemopoietic Cells to the Patients With Diagnosed Infantile Cerebral Palsy Depending on the Degrees of Compatibility of Donor and Recipient
Brief Title: Estimation of the Safety and Efficiency Transfusion of HLA Matched CBU in Patients With CP
Acronym: CP-HLA2019
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: State-Financed Health Facility "Samara Regional Medical Center Dinasty" (Other)
Collaborators: INBIO, LLC (Unknown)
Responsible Party: Principal Investigator, Volchkov Stanislav, Deputy director, Quality assurance director, State-Financed Health Facility "Samara Regional Medical Center Dinasty"
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-HLA2019
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; CP; Cord Blood; Stem cells; HLA
MeSH Terms: conditions — Cerebral Palsy | interventions — Standard of Care; Control Groups

STUDY DESIGN:
Intervention Model Description: In total, the study will involve 150 patients in three groups. The first and second groups will receive infusions of umbilical cord blood hematopoietic cells, with varying degrees of selection for the genes of the HLA system.
  The third group will be the control group. In the control group, 50 patients with similar pathology will be examined, comparable in age, sex and degree of disorder of the type of "paracopies" against the background of standard therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 Low HLA compatibility (Experimental): The patients in the first group will receive two CBU of low-level HLA matched infusions within a 6-month interval. The low-level match is 3 or less HLA compatibility degree by A, B, DRB1 loci.
  Interventions: Biological: Low HLA group CBU infusion
- Group 2 High HLA compatibility (Experimental): The patients in the second group will receive two CBU of high-level HLA matched infusions within a 6-month interval. The high-level match is 4 or more HLA compatibility degree by A, B, DRB1 loci.
  Interventions: Biological: High HLA group CBU infusion
- Standard therapy (Other): Patients with standard therapy as a control group
  Interventions: Other: Standard therapy

INTERVENTIONS:
Biological: Low HLA group CBU infusion — CB-MNC (Cord Blood Mononuclear Cells) infusion from different donors. One dose consists of 2-15х10^7 cells per 1 kg of patient weight for each infusion. The protocol includes 2 infusions with an interval of 6-x months. HLA compatibility of CB is 3 or fewer by A, B, DRB1 loci.
  Arms: Group 1 Low HLA compatibility
Biological: High HLA group CBU infusion — CB-MNC (Cord Blood Mononuclear Cells) infusion from different donors. One dose consists of 2-15х10^7 cells per 1 kg of patient weight for each infusion. The protocol includes 2 infusions with an interval of 6-x months. HLA compatibility of CB is 4 or more by A, B, DRB1 loci.
  Arms: Group 2 High HLA compatibility
Other: Standard therapy — The standard therapy can include drugs, special psychology training, etc.
  Other Names: Control group
  Arms: Standard therapy

SUMMARY:
Cerebral palsy is a disorder of movement and posture resulted from a non-progressive lesion or injury of the immature brain. It is a leading cause of childhood-onset disability.

Many experimental animal studies have revealed that umbilical cord blood is useful to repair neurological injury in the brain.

Based on many experimental studies, umbilical cord blood is suggested as a potential therapy for cerebral palsy.

This protocol was developed based on the results of the previously approved protocol of the center NCT03826498 (Allogeneic cord blood transfusion in patients with infantile cerebral palsy), which showed high efficiency in the rehabilitation of patients. The present protocol is intended for revealing the dependence of the clinical effect on the degree of tissue compatibility of umbilical cord blood samples and the recipient

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a group of neurodevelopmental conditions with abnormal movement and posture resulted from a non-progressive cerebral disturbance. It is the most common cause of motor disability in childhood. Most therapies are palliative rather than restorative. Umbilical cord blood (UCB) may be used as restorative approach for children with CP.

Many experimental animal studies have revealed that UCB is beneficial to improve and repair neurological injuries, this effect achieved due to immune regulation and angiogenesis as well as the neuroprotective effect.

Based on animal studies and some clinical trials, UCB is suggested as a potential therapy for children with CP.

This study is prospective, non randomized (open label) with control group

СLINICAL PURPOSES Estimation of the efficiency of the method of transfusion of umbilical blood hematopoietic cells to patients with diagnosed infantile cerebral palsy depending on the degrees of compatibility of donor and recipient.

RESEARCH PURPOSES

1. To develop an algorithm of using the method of transfusion of hematopoietic cells of umbilical cord blood at complex therapy of patients with children's cerebral palsy.
2. Formulate criteria for selecting patients for this method.
3. To analyze the safety and efficacy of umbilical cord blood hematopoietic cells transfusion in patients with cerebral palsy using evaluation scales.
4. To compare the efficacy of treatment of patients depending on the degree of tissue compatibility of the donor and recipient and other laboratory indications.
5. To implement the method of transfusion of umbilical cord blood hematopoietic cells in the complex therapy of patients with cerebral palsy.

ELIGIBILITY:
Patient selection criteria (indications for this type of treatment):

* Patient age from 1 to 12 years;
* Diagnosis: cerebral palsy, including postnatal damage after ischemic or hemorrhagic strokes, hypoxic or ischemic encephalopathy, periventricular leucomalacia;
* The presence of I - V lesion levels on the GMFCS - ER (CanChild) scale;
* The presence of a compatible allogeneic sample suitable for infusion;
* Parental consent (official guardians)

Patient exclusion criteria (contraindications for this type of treatment):

* Patient age up to 1 year, older than 12 years;
* The presence of the following diseases in history: heart failure in the stage of decompensation, anemia and other blood diseases;
* Decompensation of chronic and endocrinological diseases;
* Acute viral and bacterial infections during the acute clinical phase of the disease;
* HIV infection, hepatitis of B and C types;
* Oncological diseases, chemotherapy in the anamnesis;
* Tuberculosis;
* Confirmed genetic disorders;
* A severe form of intellectual disability as a concomitant disease (diagnosis can be ignored, according to the decision of the Medical Committee of the Center);
* Epileptic seizures with or without medication in the last 6 months before inclusion in the protocol.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-12-26 (Estimated); Study Completion 2024-05-26 (Estimated)

PRIMARY OUTCOMES:
Number of participants with non-serious and serious adverse events | 1 year
  Safety assessment such as adverse events will be registered. Adverse events will be monitored during all trial.
Gross Motor Function Classification System (GMFCS - ER) scale severity change | Baseline, 6 month after first infusion, 6 month after second infusion (3 times)
  Evaluation of the overall dynamics of treatment. GMFCS is a 5 level clinical classification system that describes the gross motor function of people with cerebral palsy on the basis of self-initiated movement abilities. Distinctions between levels are based on functional abilities; the need for walkers, crutches, wheelchairs, or canes/walking sticks; and to a much lesser extent, the actual quality of movement:
  Level I: Walks without Limitations Level II: Walks with Limitations Level III: Walks Using a Hand-Held Mobility Device Level IV: Self-Mobility with Limitations; May Use Powered Mobility Level V: Transported in a Manual Wheelchair The Evaluation of the results is carried out by comparing the primary and subsequent indications. Information will be collected from parents.
Changes in Standardized Gross Motor Function 66 (GMFM-66) Score for all child. | Baseline, 6 month after first infusion, 6 month after second infusion (3 times)
  GMFM (Gross Motor Function Measure) as a standardized measurement tool for assessing Gross Motor Function consisting of sub-scales; lying & rolling, sitting, crawling & kneeling, standing, walking, running & jumping (range: 0~100, a Higher value means better gross motor function). We reported changes in GMFM between each assessment time point. Categories of outcome table are baseline and values of just subtracting the latter raw scores from the former ones. This test will be acquired for all children.
Changes in The Infant Toddler Quality of Life Questionnaire for child above 3yrs. | Baseline, 6 month after first infusion, 6 month after second infusion (3 times)
  ITQOL - the 47-item short-form (ITQOL-SF47) developed for use in infants and toddlers from 2-months-to-5 years of age. Form scores physical, mental and social well being/ For each concept, item responses are scored, summed, and transformed on a scale from 0 (worst health) to 100 (best health). Changes in the completed questionnaire will be assessed. This test will be acquired for the child above 3yrs.
Changes in Ashworth scale score for all child. | Baseline, 6 month after first infusion, 6 month after second infusion (3 times)
  The Ashworth scale (AS) measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity scoring, where:
  0. No increase in tone;
  1. A slight increase in tone giving catch when the limb is moved in flexion and extension;
  2. A more marked increase in tone, but the limb is easily flexed;
  3. Considerable increases in tone, passive movement difficult;
  4. Limb rigid in flexion or extension. This test will be acquired for the child above 3yrs.

SECONDARY OUTCOMES:
Number of Participants with Chimerism (longevity) of infused cell | Baseline, 6 month after first infusion
  Chimerism study to detect the longevity of infused donor cells and predict the effectiveness of treatment. This study measures the DNA of donor cells will in patients' blood at the 6-month post-infusion. The absence of donor DNA suggests no chimerism.
The correlation between the concentration of CD14+ cells in the sample of UCB and the treatment effectiveness degree. | 1, 6 months (At each infusion)
  The correlation between the concentration of cells of the monocyte-macrophage series (CD14+) and the degree of recovery of neurological functions. Data from assessments scales with progression rate will be compared with concentration of CD14+ in infused CBU. This information will be used to assess treatment effectiveness. The assessment of a cord blood sample will be carried out on a flow cytometer immediately before the injection of the cells or in the next 12 hours.
The correlation between the concentration of CD34+ cells in the UCB and the treatment effectiveness degree | 1, 6 months (At each infusion)
  A correlation between the concentration of CD34+ cells and the degree of recovery of neurological functions. Data from assessments scales with progression rate will be compared with concentration of CD34+ cells of infused CBU. The assessment of a cord blood sample will be carried out on a flow cytometer immediately before the injection of the cells or in the next 12 hours.

CONTACTS AND LOCATIONS:
Overall Officials: STANISLAV VOLCHKOV, MD, PhD, Principal Investigator — Medical Centre Dinasty
Locations (1):
- Medical Centre Dinasty, Samara, Russia